CLINICAL TRIAL: NCT03294785
Title: Comparative Effectiveness and Cost-effectiveness of Chuna Manual Therapy for Chronic Neck Pain: A Multi-center Randomized Controlled Trial
Brief Title: Comparative Effectiveness and Cost-effectiveness of Chuna Manual Therapy for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2016-14
Record Dates: First submitted 2017-09-23; First posted 2017-09-27 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chuna manual therapy (Experimental): The Chuna manual therapy group will receive Chuna manual therapy alone. Chuna manual therapy will employ a semi-standardized treatment plan of Chuna manual therapy through Chuna technique selection based on physician judgement of techniques from Chuna Medicine (Korean Society of Chuna Manual Medicine for Spine & Nerves: Chuna Medicine: Seoul: Korean Society of Chuna Manual Medicine for Spine & Nerves; 2017) and osteopathic manipulative medicine. The Chuna techniques employed in this study are divided into cervical, thoracic and rib cage, lumbar, pelvic, sacral, pubic, and hip joint area techniques. Chuna manual therapy sessions will be administered 2 sessions/week over a period of 5 weeks (total 10 sessions). The time duration of 1 Chuna manual therapy session will consist of approximately 10-20 minutes of diagnosis and approximately 10 minutes of treatment.
  Interventions: Procedure: Chuna manual therapy
- Usual care (Active Comparator): The usual care group will receive usual care alone. Usual care will be limited to physical therapy and conventional medication in this study. Usual care will be provided with reference to a list of most frequently used treatments in neck pain-related patients from Korean Health Insurance Review and Assessment (HIRA) 2014 statistics. Frequency and types of physical therapy used will be recorded in a separate electronic case report form for outcome assessor blinding purposes.
  Interventions: Drug: Conventional medication; Procedure: Physical therapy

INTERVENTIONS:
Procedure: Chuna manual therapy — Chuna is a Korean manual therapy that has absorbed and incorporated aspects of osteopathic manipulative medicine. Chuna manual therapy utilizes spinal manipulation techniques for joint mobilization including high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement, muscle energy, and fascial techniques.
  Other Names: Chuna manipulation
  Arms: Chuna manual therapy
Drug: Conventional medication — Conventional drugs will be prescribed in an individually-tailored, pragmatic method with reference to most frequently used treatments in patients with a primary diagnosis of cervical sprain/strain group, cervical disc disorder with radiculopathy group, or cervicalgia according to Korean Health Insurance Review and Assessment (HIRA) 2014 statistics.
  Other Names: Conventional medicine; Conventional drugs
  Arms: Usual care
Procedure: Physical therapy — Physical therapy will be prescribed in an individually-tailored, pragmatic method with reference to most frequently used treatments in patients with a primary diagnosis of cervical sprain/strain group, cervical disc disorder with radiculopathy group, or cervicalgia according to Korean Health Insurance Review and Assessment (HIRA) 2014 statistics.
  Other Names: Physiotherapy
  Arms: Usual care

SUMMARY:
A multi-center randomized controlled trial assessing the comparative effectiveness and cost-effectiveness of Chuna manual therapy for chronic neck pain

DETAILED DESCRIPTION:
A multi-center randomized controlled, parallel, assessor-blinded trial will be conducted to evaluate the comparative clinical effectiveness and cost-effectiveness of Chuna manual therapy for chronic neck pain patients compared to usual care as assessed using pain, functional disability, health-related quality of life, economic evaluation, and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain patients (with pain duration of 3 months or longer)
* Patients with numeric rating scale (NRS) of radicular pain ≤ neck pain in neck pain patients with or without radiculopathy
* Patients with NRS of neck pain ≥5 during the 3 days
* Patients who have agreed to trial participation and provided written informed consent

Exclusion Criteria:

* Patients diagnosed with serious pathology(s) which may cause neck pain (e.g. spinal metastasis of tumor(s), acute fracture, spinal dislocation)
* Patients with history of neck surgery
* Patients with other chronic disease(s) which may interfere with treatment effect, safety, or interpretation of outcomes (e.g. chronic renal failure, vertebral artery complications, rheumatoid arthritis, Down syndrome)
* Patients with progressive neurologic deficit or severe neurologic symptoms such as spinal cord injury
* Patients with severe mental illness
* Patients currently taking steroids, immunosuppressants, medicine for mental illness or other medication(s) that may interfere with study results
* Patients who have received Chuna manual therapy or physical therapy, medicine such as nonsteroidal anti-inflammatory drugs (NSAIDs), or treatment(s) that may influence pain within the past week
* Pregnant patients or patients with plans of pregnancy
* Patients participating in other clinical studies or otherwise deemed unsuitable by the researchers

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Difference between visual analogue scale (VAS) of neck pain for the past 3 days at 5 weeks post-baseline and baseline | Week 5 post-baseline (screening)
  VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.

SECONDARY OUTCOMES:
Difference between visual analogue scale (VAS) of radiating arm pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6 post-baseline (screening)
  VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.
Difference between numeric rating scale (NRS) of neck pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Difference between numeric rating scale (NRS) of radiating arm pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Difference between Neck Disability Index (NDI) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The NDI evaluates functional impairment and is a 10-item questionnaire developed to assess the level of disability due to neck pain. Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to neck pain.
Difference between Northwick Park Neck Pain Questionnaire (NPQ) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The NPQ evaluates functional impairment for the past 3 days in this study and is a patient reported outcome of subjective neck pain and pain reduction. The NPQ is a 9-item questionnaire developed to assess the level of disability due to neck pain. Each item is graded into 5 levels, each representing a score of 0-4. Higher scores indicate greater limitation relating to neck pain.
Patient Global Impression of Change (PGIC) | Week 6, Month 3, 6, 9, 12 post-baseline (screening)
  PGIC grades the level of subjective improvement into 7 levels (1, very much improved; 2, much improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; and 7, very much worse).
Physical examination | Week 1, 6 post-baseline (screening)
  Pain upon movement in cervical range of motion (ROM) will be assessed.
Difference between the 5 level version of EuroQol-5 Dimension (EQ-5D-5L) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  EQ-5D is a tool developed for health-related quality of life (HRQoL) assessment, and is widely used in the health care sector. Scores range from -1, 'health worse than death' to 1, 'perfect health'. EQ-5D-5L has 5 dimensions covering current health status and functionality: mobility (M), self care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), to be rated out of 5 grades (1, no problem; 2, slight problem; 3, some/moderate problem; 4, severe problem; 5, extreme problem).
Difference between the EuroQol Visual Analogue Scale (EQ-VAS) at each timepoint and baseline, respectively | Week 1, 6 post-baseline (screening)
  EQ-VAS uses a vertical 10cm line labeled at each end with scale anchors. EQ-VAS is used to indicate the patient's health state and patients are asked to mark a point that represents their health state between the anchors of 'worst health state' and 'best health state imaginable'. Scores are recorded in millimeters with a total range of 0-100 millimeters.
Difference between the Short Form Health Survey 12 (SF-12) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  SF-12 is a simplified version of SF-36. SF-12 assesses health-related quality of life (HRQoL) across 8 domains with 1-2 items per domain: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Higher scores indicate better HRQoL.
Economic evaluation (medical costs) | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  Economic evaluation of medical costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (time-related costs) | Week 2 post-baseline (screening)
  Economic evaluation of time-related costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (lost productivity costs) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  Economic evaluation of lost productivity costs will be performed to assess cost-effectiveness of the 2 groups.
Credibility and Expectancy Questionnaire | Week 1 post-baseline (screening)
  The credibility and expectancy questionnaire will be used to assess treatment expectation on a 9-point Likert scale. Participants will be asked to select an answer to the following questions on their first visit of Week 1 (1='not at all'; and 5='somewhat'; to 9='very much'): "How much do you expect that treatment will alleviate your symptoms during the study period?"
Drug Consumption | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  Drug type and dose of prescription for medicine or rescue medicine (acetaminophen), and type and frequency of other treatments (e.g. physical therapy, injections) will be recorded.
Adverse events | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening) (every visit)
  Physicians will monitor and record any unexpected or unintended patient reaction to Chuna or usual care at each visit. Adverse events (AEs) associated with Chuna will include, but not be limited to, AEs anticipated from previous reports of manual therapy, and will stay open to all possibilities taking into consideration other potential, unknown AEs.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, MPH, Principal Investigator — Jaseng Medical Foundation
Locations (5):
- South Korea (5):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul
  - Kyung Hee University Oriental Medicine Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Cho JH, Kim KW, Lee JH, Kim MR, Kim J, Kim MY, Cho HW, Lee YJ, Lee SH, Shin JS, Prokop LL, Shin BC, Ha IH. Chuna Manual Therapy vs Usual Care for Patients With Nonspecific Chronic Neck Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2113757. doi: 10.1001/jamanetworkopen.2021.13757. PMID 34259850
- [Derived] Do HJ, Shin JS, Lee J, Lee YJ, Kim MR, Cho JH, Kim KW, Ha IH. Comparative effectiveness and economic evaluation of Chuna manual therapy for chronic neck pain: protocol for a multicenter randomized controlled trial. Trials. 2018 Nov 29;19(1):663. doi: 10.1186/s13063-018-3016-6. PMID 30497483